CLINICAL TRIAL: NCT00602056
Title: A Randomized Controlled Trial of Low Cost Interventions to Improve Adherence to Childhood Immunization Schedule in a Low Literacy Population in Pakistan
Brief Title: Low Cost Interventions to Improve Adherence to Childhood Immunization Schedule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Dr. Hussain R. Usman/Doctoral Trainee, University of Alabama at Bormingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: X050713007; X050713007
Record Dates: First submitted 2008-01-13; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Childhood Immunization Completion; Childhood Immunization Dropout; Immunization Card; Center Based Education
Keywords: Immunization dropout; Immunization card; Center based education
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Redesigned immunization card
  Interventions: Other: Redesigned immunization card
- 2 (Experimental): Center based education to mothers/caregivers
  Interventions: Other: Center based education to mothers/caregivers
- 3 (Experimental): Redesigned immunization card with center based education to mothers/caregivers
  Interventions: Other: Redesigned immunization card with center based education to mother/caregivers
- 4 (No Intervention): Standard care only

INTERVENTIONS:
Other: Redesigned immunization card — A low cost nad simplified redesigned immunization card
  Arms: 1
Other: Center based education to mothers/caregivers — A 2-3 minute center based education to mothers/caregivers
  Arms: 2
Other: Redesigned immunization card with center based education to mother/caregivers — Redesigned immunization card with center based education to mother/caregivers
  Arms: 3

SUMMARY:
The objective of the study was to assess the effect of 1) redesigned immunization card, 2) center-based education to mothers, and 3) redesigned card with center-based education to mothers, provided at DPT1, on DPT3 completion in a randomized controlled trial at rural Expanded Programme on Immunization (EPI) centers in Karachi, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All children visiting the selected EPI centers for DPT1 immunization

Exclusion Criteria:

* Not residing in the same area for last six months.

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1506 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The study outcome in each study group was the immunization status categorized into "DPT3 completed" and "DPT3 not completed". | 90 day follow-up after enrollment at DPT1 visit

CONTACTS AND LOCATIONS:
Overall Officials: Hussain R Usman, MBBS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- EPI immunization centers, Karachi, Sindh, Pakistan